CLINICAL TRIAL: NCT00355056
Title: Prospective, Randomized Investigation to Evaluate Incidence of Headache Reduction in Subjects With Migraine and PFO Using the AMPLATZER PFO Occluder to Medical Management.
Brief Title: PREMIUM Migraine Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AGA-010
Record Dates: First submitted 2006-07-19; First posted 2006-07-21 (Estimated); Results first posted 2020-07-30 (Actual); Last update posted 2020-07-30 (Actual); Status verified 2020-07

CONDITIONS: Migraine Headaches; Patent Foramen Ovale
Keywords: Migraine; PFO; Migraine Headache; patent foramen ovale
MeSH Terms: conditions — Migraine Disorders; Foramen Ovale, Patent

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Medical Management (Sham Comparator): Will not receive the closure device, and will be treated with the current standard of care medical treatment. Will undergo Intracardiac Echo (ICE) in cardiac catheterization lab and simulate PFO closure procedure (sham procedure).
  Interventions: Other: Sham Procedure
- PFO Closure (Experimental): Will undergo Intracardiac Echo (ICE) in cardiac catheterization lab and undergo PFO device closure procedure with the AMPLATZER PFO Occluder.
  Interventions: Device: AMPLATZER PFO Occluder

INTERVENTIONS:
Other: Sham Procedure — Will not receive the closure device, and will be treated with the current standard of care medical treatment. Will undergo Intracardiac Echo (ICE) in cardiac catheterization lab and simulate PFO closure procedure (sham procedure). Participants completing 1 year follow-up are eligible for PFO closure with the AMPLATZER PFO Occluder.
  Arms: Medical Management
Device: AMPLATZER PFO Occluder — Patients in this arm will receive the AMPLATZER PFO Occluder device
  Arms: PFO Closure

SUMMARY:
The Purpose of this study is to evaluate the impact of percutaneous closure of a patent foramen ovale (PFO) (a hole in the heart), using the AMPLATZER PFO Occluder, on the incidence of migraine headaches.

DETAILED DESCRIPTION:
The objective of this study is to evaluate whether percutaneous PFO closure is effective in reducing the incidence of disabling migraine headaches in patients who are refactory to medical treatment.

ELIGIBILITY:
Inclusion Criteria:

* Subjects diagnosed as having migraine headaches both with and without aura
* Have a Patent Foramen Ovale (PFO)
* A migraine history and show a refractoriness to medical treatment
* Willing to participate in follow-up visits

Exclusion Criteria:

* Subjects whose primary headaches are other than migraine headaches
* Who overuse migraine treatments
* With a clinical history of stroke or Transient Ischemic Attack (TIA)
* With contraindication to aspirin therapy and Clopidogrel
* Pregnant or desire to become pregnant within the next year

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Actual)
Dates: Start 2006-01; Primary Completion 2015-02 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sherman Sorensen, M.D., Principal Investigator — Intermountain Medical Center; Stephen Silberstein, M.D., Principal Investigator — Thomas Jefferson University; Jonathan Tobis, M.D., Principal Investigator — University of California, Los Angeles; Andrew Charles, MD, Principal Investigator — University of California, Los Angeles
Locations (30):
- United States (30):
  - St. Joseph's Hospital & Medical Center, Phoenix, Arizona
  - UCLA School of Medicine, Los Angeles, California
  - Memorial Hospital, Colorado Springs, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Medical Center of the Rockies, Fort Collins, Colorado
  - Washington Hospital Center, Washington D.C., District of Columbia
  - University of Iowa, Iowa City, Iowa
  - University of Kentucky, Lexington, Kentucky
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Tufts Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - William Beaumont Hospital, Royal Oak, Michigan
  - Abbott Northwestern Hospital, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - St. Cloud Hospital, Saint Cloud, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - St. Johns's Mercy Medical Center, St Louis, Missouri
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Children's Heart Center Las Vegas, Las Vegas, Nevada
  - Mercy Hospital of Buffalo, Buffalo, New York
  - University of Rochester Medical School, Rochester, New York
  - Pinnacle Health Hospitals, Harrisburg, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - The Methodist Hospital, Houston, Texas
  - St. Mark's Hospital, Salt Lake City, Utah
  - Intermountain Medical Center, Salt Lake City, Utah
  - Inova Healthcare Services, Falls Church, Virginia
  - University of Washington Medical Center, Seattle, Washington
  - St. Luke's Medical Center, Milwaukee, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tobis JM, Charles A, Silberstein SD, Sorensen S, Maini B, Horwitz PA, Gurley JC. Percutaneous Closure of Patent Foramen Ovale in Patients With Migraine: The PREMIUM Trial. J Am Coll Cardiol. 2017 Dec 5;70(22):2766-2774. doi: 10.1016/j.jacc.2017.09.1105. PMID 29191325

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 60 day baseline diary completion prior to randomization.
Groups:
- Sham Procedure: Did not receive the closure device, and treated with the current standard of care medical treatment.
- Patent Foramen Ovale (PFO) Device Closure: Patent foramen ovale (PFO) device Closure procedure using the AMPLATZER PFO Occluder device.
Period: Randomization Period
Arm/Group | Sham Procedure | Patent Foramen Ovale (PFO) Device Closure
Started | 107 | 123
Completed | 103 | 117
Not Completed | 4 | 6
Not completed — Early Termination | 4 | 6
Period: Optional Patent Foramen Ovale Closure
Arm/Group | Sham Procedure | Patent Foramen Ovale (PFO) Device Closure
Started | 0 (A sham procedure was not part of this period.) | 87 (Participants who completed Sham Procedure randomization Arm were eligible. 87/103 consented.)
Completed | 0 | 84
Not Completed | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Sham Procedure: Participants will not receive the closure device, and will be treated with the current standard of care medical treatment. Will undergo Intracardiac Echo (ICE) in cardiac catheterization lab and simulate PFO closure procedure (sham procedure).
- PFO Device Closure: Participants will undergo Intracardiac Echo (ICE) in cardiac catheterization lab and undergo PFO device closure procedure with the AMPLATZER PFO Occluder.
- Total: Total of all reporting groups
Arm/Group | Sham Procedure | PFO Device Closure | Total
Number analyzed (Participants) | 107 | 123 | 230
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.72 (10.16) | 42.75 (10.27) | 43.20 (10.20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 95 | 110 | 205
  Male | 12 | 13 | 25
Region of Enrollment [Number; unit: participants]
  United States | 107 | 123 | 230
International Classification of Headache Disorders (ICH) [Number; unit: participants] — Participants can have more than one International Classification of Headache Disorder, which is why the sum of the three categories exceeds the overall number of baseline participants.
  participants
    Migraine with Aura (ICH) | 71 | 80 | 151
    Migraine without Aura (ICH) | 83 | 102 | 185
    Migraine with and without Aura | 47 | 58 | 105

OUTCOME MEASURES:

1. Primary Outcome: Primary Efficacy Endpoint - Percentage of Subjects With a 50% Reduction From Baseline in the Monthly Number of Migraine Attacks at 12 Months.
Description: A 50% reduction from the monthly number of migraine attacks during the 60-day baseline phase to the monthly number of migraine attacks during month ten through the twelfth month in the treatment phase (device group versus sham group).
Time Frame: Baseline and months 10-12
Population: Participants included in the analysis were followed for 1-year, had Clinical Event Committee (CEC) adjudicated headache diaries, had greater than or equal to 60% diary compliance during the treatment phase (10-12 months) and were not treatment failures.
Measure: Number; unit: percentage of subjects
Groups:
- PFO Device Closure: PFO device Closure procedure using the AMPLATZER PFO Occluder device.
Arm/Group | Sham Procedure | PFO Device Closure
Number analyzed (Participants) | 103 | 117
percentage of subjects | 32 | 38

2. Primary Outcome: Primary Safety Endpoint - Device Related Serious Adverse Event (SAE)
Description: Number of subjects who experience a device-related major adverse event (DRMAE) through 12-months of follow-up.
  This endpoint was analyzed using an as-treated cohort that consists of all enrolled subjects who received the device (randomized and Optional PFO Closure group) and who had follow-up sufficient to adequately assess the DRMAE rate.
Time Frame: Baseline through 12 months
Population: All enrolled subjects who received the device (randomized and Optional PFO Closure group). 5 subjects were considered to have insufficient follow-up and were therefore excluded from the analysis.
Measure: Number (99% Confidence Interval); unit: percentage of participants
Arm/Group | PFO Device Closure
Number analyzed (Participants) | 205
percentage of participants | 0.49 [0.01 to 2.69]

3. Secondary Outcome: Change in Mean Migraine Days/Month
Description: Change in the number of migraine days is calculated by the difference in the mean number of migraine days between the baseline assessment period and the treatment phase (months 10-12 post-procedure) for the respective randomization groups.
Time Frame: Baseline and months 10-12
Measure: Mean (Standard Deviation); unit: Migraine days per month
Groups:
- Sham Procedure: Sham Procedure and treated only with current standard of care medical treatment.
- PFO Device Closure: Patients in this arm received the AMPLATZER PFO Occluder device
Arm/Group | Sham Procedure | PFO Device Closure
Number analyzed (Participants) | 103 | 117
Migraine days per month | 2.0 (5.0) | 3.4 (4.4)

4. Secondary Outcome: Percentage of Subjects With Successful PFO Closure at 12-months
Description: Successful Closure by Core Lab Adjudicated Transcranial Doppler (TCD) Grade <= 2
Time Frame: Baseline and month 12
Population: 117 device subjects completed the 12 month visit. Only 104 had TCDs that were able to be adjudicated. Of the 13 device subjects with unadjudicated TCDs, 4 did not have valsalva data and 9 did not have TCD data available for various reasons.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- PFO Closure: Device group subjects who had a Core Lab adjudicated TCD grade at Valsalva of less than or equal to 2 at 12-months.
Arm/Group | PFO Closure
Number analyzed (Participants) | 104
percentage of participants | 82.7 [74 to 89]

5. Secondary Outcome: Change in Migraine Disability Assessment (MIDAS) Score From Baseline to 12-months
Description: The MIDAS questionnaire measure the impact of headaches on daily living. A total score of 0-5 equals little to no disability, 6-10 equals mild disability, 11-20 equals moderate disability, and a score 21 or greater equals severe disability. The maximum possible score is 276.
Time Frame: 12 months
Population: 101 participants in the sham group and 116 subjects in the PFO device closure group had both baseline and 12-month MIDAS scores available to perform the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sham Procedure | PFO Device Closure
Number analyzed (Participants) | 101 | 116
units on a scale | -17 (36) | -22.6 (32.9)

6. Secondary Outcome: Incidence of a 75% Reduction in Migraine Headache Attacks
Time Frame: 12 months
Population: Participants were included in the analysis were followed for 1-year, have CEC adjudicated headache diaries, had greater than or equal to 60% diary compliance during the treatment phase (10-12 months) and were not treatment failures.
Measure: Number; unit: percentage of participants
Arm/Group | Sham Procedure | PFO Device Closure
Number analyzed (Participants) | 103 | 117
percentage of participants | 16.5 | 20.5

7. Secondary Outcome: Procedural Success
Description: Procedural success is calculated by the percent of device group subjects who were implanted with the study device and experienced no serious device or procedure-related adverse events.
Time Frame: 12 months
Population: Device group subjects who were implanted with the study device and experienced no serious device or procedure-related adverse events.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | PFO Closure
Number analyzed (Participants) | 123
percentage of participants | 94.3 [88.6 to 97.7]

8. Secondary Outcome: Long-Term Success
Description: Percent of PFO closure group subjects who were implanted with the study device, experienced no serious device or procedure-related adverse events and have a core-lab adjudicated TCD Grade at Valsalva ≤ 2 at 1-year.
Time Frame: 12 months
Population: Percent of PFO closure group subjects who were implanted with the study device, experienced no serious device or procedure-related adverse events and have a core-lab adjudicated TCD Grade at Valsalva ≤ 2 at 1-year. 117 device subjects completed the 12 month visit. Only 104 had TCDs that were able to be adjudicated.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | PFO Closure
Number analyzed (Participants) | 104
percentage of participants | 80.8 [71.9 to 87.8]

9. Secondary Outcome: Incidence of All Adverse Events at 12-months
Time Frame: 12 months
Population: Participants who experienced an adverse event at or before 12-months post-procedure
Measure: Number; unit: participants
Arm/Group | Sham Procedure | PFO Device Closure
Number analyzed (Participants) | 107 | 123
participants | 93 | 105

10. Secondary Outcome: Incidence of Device-related Adverse Events
Time Frame: 12 months
Population: Participants who experienced a device-related adverse event, as adjudicated by the Data Safety and Monitoring Board (DSMB), at or before 12-months post-procedure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | PFO Closure
Number analyzed (Participants) | 123
percentage of participants | 31.7 [23.6 to 40.7]

11. Secondary Outcome: Incidence of a 95% Reduction in Migraine Headache Attacks
Time Frame: 12-months
Measure: Number; unit: percentage of participants
Arm/Group | Sham Procedure | PFO Device Closure
Number analyzed (Participants) | 103 | 117
percentage of participants | 0.97 | 8.55

12. Other Pre Specified Outcome: Change in Beck Depression Inventory (BDI) Scale
Description: The difference in BDI between baseline and 12-months for the respective randomization groups. The highest possible score of the BDI is 63, which represents extreme depression. The lowest possible score is 0, which represents no depression.
Time Frame: 12 months
Population: 101 participants in the sham group and 116 subjects in the PFO device closure group had both baseline and 12-month BDI scores available to perform the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sham Procedure | PFO Device Closure
Number analyzed (Participants) | 101 | 116
units on a scale | -0.3 (7.1) | -2.1 (6.5)

13. Post Hoc Outcome: Responder Rate for Subjects in Whom Majority of Attacks Were With Aura
Description: The term "majority" in "majority of migraine attacks included aura" was defined by the Neurologist (>50%) at the time of randomization based on a review of the subject's study baseline headache diary and medical history.
Time Frame: 12 months
Measure: Number; unit: percentage of subjects
Arm/Group | PFO Device Closure | Sham Procedure
Number analyzed (Participants) | 39 | 40
percentage of subjects | 48.7 | 22.5

14. Post Hoc Outcome: Percentage of Subjects With Migraine With Aura Determined to Have a Complete Cessation of Migraine Attacks According to the International Headache Society (IHS)
Description: Complete Cessation of Migraine Attacks, baseline diary compared to months 10-12
Time Frame: Baseline through months 10-12
Population: 6 PFO Device Closure Subjects and 3 Sham Procedure Subjects with Aura do not have 12-month follow-up data available.
Measure: Number; unit: percentage of subjects
Arm/Group | PFO Device Closure | Sham Procedure
Number analyzed (Participants) | 74 | 68
percentage of subjects | 10.8 | 1.5

ADVERSE EVENTS:
Time Frame: All adverse events were collected from the time of signing informed consent until the 12-month follow-up visit. After the 12-month follow-up visit, serious adverse events and/or device-related events were collected until completion of study requirements.
Groups:
- Optional PFO Closure: Subjects randomized to the sham arm and completed their 12-month follow up visit were given the option of PFO closure with the Amplatzer PFO Occluder.
Arm/Group | PFO Device Closure | Sham Procedure | Optional PFO Closure
Serious Adverse Events (participants affected / at risk) | 1/123 | 0/107 | 0/87
Other Adverse Events (participants affected / at risk) | 119/123 | 103/107 | 68/87
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PFO Device Closure (N=123) | Sham Procedure (N=107) | Optional PFO Closure (N=87)
Transient atrial fibrillation after device placement (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PFO Device Closure (N=123) | Sham Procedure (N=107) | Optional PFO Closure (N=87)
Arterial Hypertension/Hypertension (Cardiac disorders) | 8 (9) | 4 (4) | 2 (2)
Nausea (General disorders) | 10 (11) | 9 (9) | 1 (1)
Fatigue/Generalized Fatigue (General disorders) | 4 (5) | 10 (11) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 8 (9) | 4 (4) | 0 (0)
Musculoskeletal Pain (General disorders) | 21 (22) | 9 (10) | 0 (0)
Common cold/Upper Respiratory Tract Infection (Infections and infestations) | 29 (35) | 28 (39) | 3 (3)
Abdominal Pain (Gastrointestinal disorders) | 17 (18) | 14 (14) | 1 (1)
Anxiety (General disorders) | 7 (7) | 5 (5) | 1 (1)
Rash (General disorders) | 10 (11) | 4 (4) | 1 (1)
Pain (General disorders) | 7 (9) | 8 (9) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 16 (17) | 13 (15) | 4 (4)
Diarrhea (Gastrointestinal disorders) | 7 (7) | 4 (4) | 0 (0)
Dizziness (General disorders) | 6 (6) | 9 (12) | 2 (2)
Palpitations (Cardiac disorders) | 30 (31) | 16 (18) | 12 (12)
Sinusitis (General disorders) | 29 (35) | 23 (40) | 7 (7)
Chest Pain (General disorders) | 22 (28) | 13 (13) | 13 (13)
Vascular Access Site Complication Pain (Vascular disorders) | 22 (22) | 12 (13) | 9 (9)
Bruise/Purpura Simplex (General disorders) | 20 (21) | 27 (31) | 10 (10)
Viral Syndrome (General disorders) | 9 (9) | 3 (5) | 0 (0)
Low Back Pain (General disorders) | 7 (8) | 3 (3) | 1 (1)
Back Pain (General disorders) | 8 (8) | 11 (12) | 5 (5)
Vascular Access Site Complication Hematoma (Vascular disorders) | 8 (8) | 12 (12) | 6 (6)
Vascular Access Site Complication Bruise (Vascular disorders) | 8 (8) | 3 (3) | 3 (3)
Mid-Sternal Chest Pressure (General disorders) | 6 (7) | 0 (0) | 1 (1)
Headache (General disorders) | 6 (6) | 7 (7) | 2 (2)
Depression (General disorders) | 3 (3) | 6 (7) | 1 (1)
Dyspnea (General disorders) | 6 (6) | 7 (7) | 2 (2)
Sore Throat (General disorders) | 4 (5) | 7 (7) | 1 (1)
Vascular Access Site Complication Bleeding (Vascular disorders) | 5 (5) | 3 (3) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other